CLINICAL TRIAL: NCT04740320
Title: Screening Protocol for a Dose Finding Human Experimental Infection Study in Healthy Subjects Using a GMP-produced SARS-COV-2 Wild Type Strain
Brief Title: COVID-19 SARS-CoV-2 Screening Protocol
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Hvivo (Industry)
Responsible Party: Sponsor
Other Study IDs: 20IC6378
Record Dates: First submitted 2021-01-26; First posted 2021-02-05 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Covid19
Keywords: COVID19; Coronavirus; Coronavirus disease 19; SARS-COV-2; Healthy volunteer; human challenge
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — Samples of tissue, cells and fluids will be stored according to Imperial College London and hVIVO SOPs as appropriate. Samples will be pseudoanonymised with participant identification numbers only and the anonymisation key kept in a separate locked location accessible only to the hVIVO clinical study team. Samples may be used for further assays or in other ethically approved studies. Samples and data may be shared with UK and international collaborators in studies that have been approved by local ethics committees and subject to a valid Materials Transfer Agreement. At the end of the study any remaining samples will be either destroyed, transferred to the sponsor or subject to consent, transfer to and maintained under hVIVOs HTA licenses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Volunteers asked to register details on a SARS-CoV-2 specific web page UKcovidchallenge.com. They will be contacted with a short webform questionnaire to be performed prior to a follow-up telephone questionnaire or will be asked to complete a telephone questionnaire. If inclusion/exclusion criteria are met, appointment for a screening visit will be scheduled. Screening appointments will be conducted at hVIVO. Written consent for screening will be obtained prior to any history-taking, examination or tests are carried out. Medical history will be requested from GP to assess suitability. Once the SARS-CoV-2 characterization study is approved, potential participants will be given the study specific PIS detailing the full study and experimental procedures. The opportunity to discuss further and ask questions will be available prior to booking a study visit.

SUMMARY:
The aim of this screening protocol is to assess volunteers for their potential eligibility to participate in a dose finding human experimental infection study in healthy subjects using a GMP-produced SARS-CoV-2 wild type strain

DETAILED DESCRIPTION:
Recruitment will be done through a number of channels:

* Approved advertising, including social medial
* hVIVO volunteer database
* Referral
* Organic search, i.e. where the volunteer has learned of this study by doing a Google search or through friends or family rather than due to any advertising Following Research Ethics Committee approval of the full study, screened subjects who confirm their willingness to participate in the SARS-CoV-2 human infection challenge characterization study will be invited to consider the study-specific PIS-ICF and enter the final study consenting process.

The number of subjects who are to be recruited will depend on specific sample-size requirements for the SARS-CoV-2 human infection characterization study.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent document signed and dated by the participant and the Investigator.
2. Male or female, age between 18 and 30 years inclusive (at the time of the study consent)
3. Seronegative to the challenge virus SARS-CoV-2
4. Women of childbearing potential with a documented menstrual period within 28 days before the first dose (unless using a contraceptive method that suppressed menstruation as indicated in the study protocol) and willing and able to use contraception as described in the study protocol from 4 weeks before the scheduled date of viral challenge until 30 days after receipt of the final dose of study medication. Negative urine pregnancy test will be required at screening plus, on admission to the quarantine unit, a Negative serum beta human chorionic gonadotropin (β-hCG) is a required. Also a negative urinary pregnancy test prior to virus challenge is also required.
5. Men who are willing to use one of the contraception methods described in the study protocol, from the time of the date of viral challenge, until 90 days after receipt of the final dose of study medication.
6. In good health with no history of clinically significant medical conditions (as described in Exclusion criteria) that would interfere with subject safety, as defined by medical history, physical examination and routine laboratory tests, ECG, and Chest X-Ray* and determined by the Investigator at a screening evaluation and/or at admission to the Quarantine Unit.
7. Subjects will have a documented medical history either prior to entering the study and/or following medical history review with the study physician at screening
8. Using the QCOVID tool, an absolute risk of COVID-associated death of 1 in 250,000 (0.0004%) or less and COVID-associated hospital admission of 1 in 5000 (0.02%) or less), or alternative risk threshold at the discretion of the CI with advice from the DSMB

   Exclusion Criteria:

   Any potential subject who meet any of the criteria below will be excluded from participating in this study.

   Clinical history 1. History or evidence of any clinically significant or currently active cardiovascular, (including thromboembolic events), respiratory, dermatological, gastrointestinal, endocrine, haematological, hepatic, immunological, rheumatological, metabolic, urological, renal, neurological, psychiatric illness. Specifically:

   a) Subjects with any history of physician diagnosed and/or objective test confirmed asthma, chronic obstructive pulmonary disease, pulmonary hypertension, reactive airway disease, or chronic lung condition of any aetiology or who have experienced:

   o Significant/severe wheeze in the past
   * Respiratory symptoms including wheeze which has ever resulted in hospitalisation
   * Known bronchial hyperreactivity to viruses b) History of thromboembolic, cardiovascular or cerebrovascular disease c) History or evidence of diabetes mellitus d) Any concurrent serious illness including history of malignancy that could interfere with the aims of the study or a subject completing the study. Basal cell carcinoma within 5 years of treatment or with evidence of recurrence is also an exclusion e) Migraine with associated neurological symptoms such as hemiplegia or vision loss. Cluster headache/migraine or prophylactic treatment for migraine f) History or evidence of autoimmune disease or known immunodeficiency of any cause.

     g) Other major disease that, in the opinion of the Investigator, could interfere with a subject completing the study and necessary investigations.

     h) Immunosuppression of any type. 2. Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx, a clinically significant history of epistaxis (large nosebleeds) within the last 3 months, nasal or sinus surgery within 6 months of inoculation.

     3. Clinically active rhinitis (including hay fever) or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine.

     4. History of anaphylaxis and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the PI.

     5. History or presence of alcohol addiction, or excessive use of alcohol (average weekly intake in excess of 28 units alcohol; one unit being a half glass of beer, a small glass of wine or a measure of spirits).

     6. Psychiatric illness including subjects with a history of depression and/or anxiety with associated severe psychiatric comorbidities, for example psychosis. Specifically,

     a) Subjects with history of anxiety-related symptoms of any severity within the last 2 years if the Generalized Anxiety Disorder-7 score is ≥4 b) Subjects with a history of depression of any severity within the last 2 years if the Patient Health Questionnaire-9 score is ≥4

     7. Current smokers or subjects who have smoked ≥5 pack years at any time [5 pack years is equivalent to one pack of 20 cigarettes a day for 5 years].

     • Subjects who have smoked <5 pack years - at any time in the 3 months prior to admission to the quarantine unit they have used tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch) or electronic cigarettes.

     8. Family history of 1st degree relative aged 50 years or less with sudden cardiac or unexplained death 9. Family History of Severe COVID or response to any other viral disease e.g. Guillain-Barré Measurements and investigations
     1. A total body weight of ≤ 50g and a Body Mass Index (BMI) ≤18 kg/m2 and ≥28 kg/m2. The upper limit of BMI may be increased to ≤ 30kg/m2 at the PI's discretion, in the case of physically fit muscular individual
     2. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
     3. Any clinically significant abnormal finding on screening biochemistry, haematology and microbiology blood tests or urinalysis i.e. grade 1 lab abnormalities (or above, see Appendix 4 Toxicity Grading Scale for Laboratory AEs) apart from minor deviations which are clinically acceptable and approved by the Principal Investigator

        a) Elevated random glucose and HbA1C b) Positive HIV, active/chronic hepatitis A, B or C test. c) Confirmed positive test for drugs of abuse on admission and urinary cotinine at quarantine.
     4. A forced expiratory volume in 1 second (FEV1) and a forced vital capacity (FVC) <80% of predicted value calculated using ATS/ERS guidance
     5. Twelve-lead ECG recording with clinically relevant abnormalities as judged by the study physician/PI.

        Recent respiratory infection
     6. History of, or currently active symptoms suggestive of upper or lower respiratory tract infection (including reduced sense of taste and smell, raised body temperature and/or persistent cough) within 6 weeks prior to viral challenge.
     7. Presence of cold-like symptoms and/or fever (defined as subject presenting with a temperature reading of >37.9ºC) Receipt of medications and interventions
     8. Evidence of a live vaccine within 60 days prior to the planned date of viral challenge, a non-live vaccine within 30 days prior to the planned date of viral challenge, or intention to receive any vaccination(s) before the day 28 follow-up visit. (NB. No travel restrictions applied after the Day 28 Follow-up visit).
     9. Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned date of viral challenge or planned during the 3 months after the final visit.
     10. Medications

         a) Use of any medication or product (prescription or over-the-counter), for symptoms of hayfever, nasal congestion or respiratory tract infections or dermatitis/eczema including the use of regular nasal or medium-high potency dermal corticosteroids, antibiotics and First Defence™ (or generic equivalents) within 7 days prior to the planned date of viral challenge apart from those described and allowed in Permitted Medication or agreed by the Principle Investigator b) Receipt of any investigational drug within 3 months prior to the planned date of viral challenge.

         c) Receipt of three or more investigational drugs within the previous 12 months prior to the planned date of viral challenge.

         d) Prior inoculation with a virus from the same virus-family as the challenge virus.

         e) Receipt of systemic (intravenous and/or oral) glucocorticoids or systemic antiviral drugs within 6 months prior to the planned date of viral challenge.

         f) Over the counter medications (e.g., paracetamol or ibuprofen) where the dose taken over the preceding 7 days prior to the planned date of viral challenge had exceeded the maximum permissible 24-hour dose (e.g., >4g per day of paracetamol over the preceding week).

         g) Use or anticipated use within 7 days prior to the planned date of viral challenge and during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows.

         h) Chronically used medications, vitamins or dietary supplements, including any medication known to be a moderate/potent inducer or inhibitor of cytochrome P450 enzymes, within 21 days prior to the planned date of viral challenge.

         i) Subjects who have received any systemic chemotherapy agent, immunoglobulins, or other cytotoxic or immunosuppressive drugs at any time.
     11. Prior participation in another human viral challenge study in the preceding 12 months taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study.
     12. Any nasal sampling procedure in the 6 months before date of expected viral challenge in this study. Nasal swabs are allowed.

         General
     13. Subject was mentally or legally incapacitated in the opinion of the Investigator.
     14. Females who:

         1. Are breastfeeding within 6 months of study commencement, or
         2. Had been pregnant within 6 months prior to the study, or
         3. Had a positive pregnancy test at any point during screening or prior to inoculation with challenge virus
     15. Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 3 years, the elderly (>65 years), immunosuppressed persons, or those with chronic respiratory disease Other
     16. Was employed or was a first-degree relative of anyone employed by the Sponsor, a participating clinical trial site, or any Contract Research Organisation involved in the study.
     17. Any other reason that the Investigator considered made the subject unsuitable to participate.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers aged 18-30
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Chiu, Principal Investigator — Imperial College London
Locations (1):
- hVIVO Services Ltd, QMB Bioenterprise building, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Geometric Mean (Standard Deviation); unit: age of participants] | 21.8 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 36

OUTCOME MEASURES:

1. Primary Outcome: Participants Enrolled
Description: Number of participants enrolled in main study
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
Participants | 36

ADVERSE EVENTS:
Time Frame: N/A This is a screening protocol and Adverse Events are not captured as part of this.
Description: N/A This is a screening protocol and Adverse Events are not captured as part of this.
Arm/Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT04740320/Prot_000.pdf